CLINICAL TRIAL: NCT06895876
Title: Deep Parasternal Intercostal Plane Block : Effect on the Quality of Postoperative Recovery After Cardiac Surgery
Brief Title: Deep Parasternal Intercostal Plane Block
Acronym: DPIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute Arnault Tzanck, France (Other)
Responsible Party: Principal Investigator, Marc LOPEZ, MD, Investigator principal, Institute Arnault Tzanck, France
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-A01183-38
Record Dates: First submitted 2022-03-04; First posted 2025-03-26 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Nerve Block
Keywords: Transversus thoracic muscle plane block; Cardiac surgery; Postoperative analgesia; Quality of recovery; QoR-15

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deep parasternal intercostal plane block (Experimental): The block is performed bilaterally in the 4th intercostal space. The probe is placed in the latero-median axis and a needle is placed latero-medially between the intercostal and transverse thoracic muscle. The solution is then injected under ultrasound control ()20 mL of 0,375% Naropeïne
  Interventions: Procedure: Deep parasternal intercostal plane block
- Control (No Intervention): Standard multimodal analgesia

INTERVENTIONS:
Procedure: Deep parasternal intercostal plane block — The block is performed bilaterally in the 4th intercostal space. The probe is placed in the latero-median axis and a needle is placed latero-medially between the intercostal and transverse thoracic muscle. The solution is then injected under ultrasound control
  Arms: Deep parasternal intercostal plane block

SUMMARY:
Cardiac surgery is a source of severe post operative pain witch can cause major respiratory complications due to non optimal post operative rehabilitation.

Multimodal analgesia provides acceptable pain control , but does not seem sufficient during coughing or mobilization. The use of morphine also exposes patients to side effects (nausea, vomiting, pruritus, respiratory depression, chronic pain, ileus). Bleeding and hemodynamic risks of peridural and spinal aneshesia limits their use.

The postoperative efficacy of deep parasternal intercostal plane block has not yet been evaluated sufficiently. The aim of this study is to evaluate the efficacity of TTMPB on the quality of postoperative recovery after cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring cardiac surgery with sternotomy

Exclusion Criteria:

* Emergency procedure
* Procedures requiring lateral chest drainage
* Hemodynamic instability
* Severe kidney or liver failure
* BMI > 40
* Chronic pain
* Allergy to local anesthesics
* Pregnant woman
* Long term opioïds use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2022-08-10 (Actual); Primary Completion 2025-02-12 (Actual); Study Completion 2025-06-15 (Actual)

PRIMARY OUTCOMES:
Quality of recovery 15 (QoR-15) | 24 hours after surgery
  QoR-15 score : 0 to 150. Addition of 15 items note between 0 to 10 150 = perfect post operative recovery possible 0 = worst post operative recovery possible

SECONDARY OUTCOMES:
Total morphine consumption at 24 hours | 24 hours after surgery
  Total morphine consumption, in milligrams, during the first 24 hours after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Arnault Tzanck, Saint-Laurent-du-Var, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kehlet H. Multimodal approach to control postoperative pathophysiology and rehabilitation. Br J Anaesth. 1997 May;78(5):606-17. doi: 10.1093/bja/78.5.606. PMID 9175983
- [Background] Mangano DT, Siliciano D, Hollenberg M, Leung JM, Browner WS, Goehner P, Merrick S, Verrier E. Postoperative myocardial ischemia. Therapeutic trials using intensive analgesia following surgery. The Study of Perioperative Ischemia (SPI) Research Group. Anesthesiology. 1992 Mar;76(3):342-53. PMID 1531742
- [Background] Aydin ME, Ahiskalioglu A, Ates I, Tor IH, Borulu F, Erguney OD, Celik M, Dogan N. Efficacy of Ultrasound-Guided Transversus Thoracic Muscle Plane Block on Postoperative Opioid Consumption After Cardiac Surgery: A Prospective, Randomized, Double-Blind Study. J Cardiothorac Vasc Anesth. 2020 Nov;34(11):2996-3003. doi: 10.1053/j.jvca.2020.06.044. Epub 2020 Jun 18. PMID 32665179